CLINICAL TRIAL: NCT03633253
Title: The "Motoric Cognitive Risk" Syndrome in the Quebec Population: Results From the NuAge Study
Brief Title: The "Motoric Cognitive Risk" Syndrome in the Quebec Population
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: CODIM-FLP-16 288
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cognition Disorders in Old Age; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCR syndroms
  Interventions: Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages
- Non MCR syndroms
  Interventions: Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages

INTERVENTIONS:
Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages — First, prevalence of MCR syndrome will be determined by classifying participants into MCR and non-MCR syndrome groups. Second, between-group comparisons of participants' characteristics will be performed using unpaired t-test, Mann-Whitney, analysis of variance with LSD correction or Chi-square test, as appropriate. Third, multiple regressions will be performed to examine the association between MCR syndrome (dependent variable) and cardio-vascular risk factors and/or diseases (independent variables) adjusted on participants' characteristics. Fourth, the incidence of MCR syndrome during the follow-up period of NuAge study will be reported. Fifth, regression will be performed to examine the association between MCR syndrome (dependent variable) and cognitive decline as well cognitive impairment (independent variables, separated model) adjusted on participants' characteristics.

SUMMARY:
The overall objective of the proposal is to examine the epidemiology of the newly reported "motoric cognitive risk" (MCR) syndrome, which is a pre-dementia syndrome combining subjective cognitive complaint (i.e.; memory complaint) with objective slow gait speed, in the Quebec elderly population.

Cognition and locomotion are two human abilities controlled by the brain. Their decline is highly prevalent with physiological and pathological aging, and is greater than the simple sum of their respective prevalence, suggesting a complex age-related interplay between cognition and locomotion. Both declines in cognition and locomotion are associated, furthermore the temporal nature of their association has been unclear for a long time. Recently, a systematic review and meta-analysis has provided evidence that poor gait performance predicts dementia and, in particular, has demonstrated that MCR syndrome is a pre-dementia syndrome, suggesting that low gait performance is the first symptom of dementia. The uniqueness of MCR syndrome is that it does not rely on a complex evaluation or laboratory investigations. Indeed, this syndrome combined subjective cognitive complaint and objective slow gait speed, and is easy to apply in population-based settings.

Prevalence and incidence of MCR syndrome, as well as its association with incidence of cognitive decline and impairment, have never been reported in Canada. Nutrition as a determinant of successful aging: The Quebec longitudinal Study (the NuAge study) is a Quebec population-based observational cohort study performed in healthy older community-dwellers adults which provides a unique opportunity to: 1) obtain reliable estimates of MCR syndrome prevalence and incidence, 2) determine the distribution of clinical characteristics associated with MCR syndrome, 3) examine the association of MCR syndrome with cognitive decline and incidence of cognitive impairment in the Quebec elderly population.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for this study will be participants of the NuAge study

Exclusion Criteria:

Individuals not eligible for the NuAge study, No information about cognitive complaint, No measure of walking speed, No follow-up completed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals eligible for this study will be participants of the NuAge study (n=1,793). All included participants of NuAge Study were healthy and, in particular, they were cognitively intact at baseline and had no mobility disability.
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
MCR syndrome criteria | 1 day
  Diagnosis of MCR syndrome following Verghese et al. criteria

SECONDARY OUTCOMES:
Cognitive decline and impairment | 1 day
  Modified Mini-Mental State (3MS) in the NuAge study.
Covariates | 1 day
  Cardio-vascular risk factors and diseases assessed using reported health condition
Covariates | 1 day
  Cardio-vascular risk factors and diseases assessed using physical examination: body mass index
Covariates | 1 day
  Cardio-vascular risk factors and diseases assessed using physical examination: hip waist ratio from hip and waist circumference
Covariates | 1 day
  Cardio-vascular risk factors and diseases assessed using physical examination: blood pressure (value of systolic, diastolic when participants are seated in an upright position in a chair)

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No